CLINICAL TRIAL: NCT01730599
Title: A Longitudinal 5 Years Follow up Study in Parkinson's Disease (PD) Patients Carriers of the LRRK2 Gene G2019S Mutation
Brief Title: A Longitudinal Study in Parkinson's Disease (PD) Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-11-NG-0473
Record Dates: First submitted 2012-10-22; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PD patients: PD patients carriers of the G2019S mutation in the LRRK2 gene
  Interventions: Other: neurological exam

INTERVENTIONS:
Other: neurological exam — motor and cognitive functions

SUMMARY:
This is a longitudinal study in patients with Parkinson's Disease (PD) carriers of a genetic mutation - substitution of gly with ser in position 2019 (G2019S) in the leucine-rich repeat kinase 2 (LRRK2) gene. The purpose of this study is to explore the association between genetic mutations in the known genes and their influence on disease manifestation over few years of follow up

ELIGIBILITY:
Inclusion Criteria:

* parkinson'd disease patients that already participated in a pasr cross sectional study

Exclusion Criteria:

* subjects with cognitive decline by the parameters defined in Diagnostic and Statistical Manual of Mental Disorders (DSM)- IV
* subjects with psychiatric disorder
* subjects unable to sign a consent form

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients carriers of the G2019S mutation in the LRRK2 gene
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
change from baseline in updrs motor and total scores | the participants will be followed for 5 years. the measurements will be taken evry 18 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel